CLINICAL TRIAL: NCT05032339
Title: Evaluation of the Plasma Cell Disorders Panel (BD OneFlow™ PCST and BD OneFlow™ PCD) on the BD FACSLyric™ Flow Cytometer Using Leftover, De-identified Specimens
Brief Title: Evaluation of the Plasma Cell Disorders Panel on the BD FACSLyric™ Flow Cytometer
Status: Completed | Type: Observational
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: CAS-OFLYRICPP-IVDR
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Plasma Cell Disorder
Keywords: leukemia & lymphoma
MeSH Terms: conditions — Neoplasms, Plasma Cell; Leukemia; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Remnant/ Leftover specimens: Specimens that meet inclusion/exclusions criteria and are leftover from routine flow cytometry testing for plasma cell disorders
  Interventions: Diagnostic Test: IUO Plasma Cell Disorders Panel

INTERVENTIONS:
Diagnostic Test: IUO Plasma Cell Disorders Panel — This Investigational Panel , comprised of 2 reagents , is intended for in vitro diagnostic use for qualitative flow-cytometric immunophenotyping of plasma cell populations. These reagents are used as an aid in the differential diagnosis of hematologically abnormal patients having, or suspected of having, plasma cell disorders.

SUMMARY:
Multi-site, prospective performance study to determine equivalency between the investigational OneFlow PCD panel on the FACSLyric system versus the final clinical diagnosis.

DETAILED DESCRIPTION:
Hematology laboratories rely on flow cytometry technology (in addition to classic hematological methods) to aid in screening, diagnosing, and monitoring patients with hematological disorders. High speed and broad applicability of flow cytometry allows for the diagnosis and accurate focus on targets. Currently, there are no general consensus panels being used; as a consequence, the leukemia & lymphoma (L&L) testing remains a single-vial antibody being used, with various in-house laboratory developed tests (LDTs) being used to test patient specimens. Furthermore, the analysis of flow cytometer generated data is not standardized and requires a high level of expertise/training for interpretation of complex data. Therefore, optimized and standardized immunostaining protocols for the diagnosis, classification, and prognostic sub-classification of hematological malignancies are needed.

This Investigational panel for plasma cell disorders is intended for in vitro diagnostic use for qualitative flow-cytometric immunophenotyping of plasma cell populations on the BD FACSLyric flow cytometer. These reagents are used as an aid in the differential diagnosis of hematologically abnormal patients having, or suspected of having, plasma cell disorders.

Enrollment will occur at up to 8 investigational sites . Data will be acquired from Eligible remnant/leftover specimens on the BD FACSLyric flow cytometer and evaluated by site personnel and expert analysts .

The final diagnosis and the affected cell population will be determined by site standard of care .

Analysis of data will evaluate identification of normal vs abnormal cell population of the expert & site analysts as compared to the final diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Specimen collected/handled prior to enrollment in accordance with site policies and procedures.
2. Specimen with adequate volume (approximately 300 µL) to complete protocol tests.
3. Specimen is leftover BM from routine flow cytometry laboratory testing for plasma cell disorders, other hematological disorders, non-hematological tumors, and other hematological disorders (non-malignant).
4. Specimen from a newly diagnosed or relapsed subject.
5. Specimen is stored at room temperature, upon receipt by the site.
6. Age of specimen (time of collection to start of first pre-wash): ≤24 hours.
7. Specimen collected in EDTA (K2 or K3) or heparin (sodium or lithium).
8. Specimens are from subjects irrespective of race, gender, and ethnicity.

Exclusion Criteria:

1. Specimen from healthy subject.
2. Specimen from subject <22 years old.
3. Specimen from subject undergoing any treatment for any form of L&L.
4. Specimen from subject with minimal residual disease (MRD) as determined by site.
5. Visibly clotted specimen.
6. Visibly hemolyzed specimen.
7. Frozen specimen.
8. Refrigerated specimen.
9. Fixed specimen.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A minimum of 150 remnant/leftover bone marrow specimens from routine flow cytometry laboratory testing for plasma cell disorders, other hematological disorders, non-hematological tumors, and other hematological disorders (non-malignant). Specimens from healthy subjects will be excluded.
  At least 75 specimens must have abnormal plasma cells, at least 75 must have normal polyclonal plasma cells.
  Specimens are from subjects irrespective of race, gender, and ethnicity. Subjects above 22 years of age
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Comparison between expert analysts' determination of normal and abnormal specimen and final diagnosis | Age of specimen for Peripheral Blood (PB) andBone Marrow (BM) (time of collection to start of first pre-wash): ≤ 24 hours.
  Determine equivalence between the investigational OneFlow PCD Panel on FACSLyric system results analyzed by two independent experts versus the final clinical diagnosis for normal polyclonal plasma cells or abnormal plasma cells using leftover, hematologically abnormal specimens.
  Sensitivity and specificity will be calculated .

CONTACTS AND LOCATIONS:
Overall Officials: Imelda Omana-Zapata, MD, PHD, Study Director — Becton, Dickinson and Company
Locations (5):
- Corepath Laboratories, San Antonio, Texas, United States
- Champalimaud Foundation, Lisbon, Portugal
- University of Salamanca, Salamanca, Spain
- Kantonsspital Aarau, Aarau, Switzerland
- Cambridge university hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No